CLINICAL TRIAL: NCT01339507
Title: A Patient Reported Ocular Comfort Assessment Comparing Bepreve to Lastacaft in Patients With a History of Allergic Conjunctivitis
Brief Title: A Patient Reported Ocular Comfort Assessment Comparing Bepreve to Lastacaft
Status: Completed | Type: Observational
Sponsor: Cunningham, Derek N., O.D., P.A. (Individual)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Principal Investigator, Derek N. Cunningham, PI, Cunningham, Derek N., O.D., P.A.
Other Study IDs: MAC-05-11
Record Dates: First submitted 2011-04-19; First posted 2011-04-20 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Bepreve: Subjects with a history of allergic conjunctivitis.
- Lastacaft: Subjects with a history of allergic conjunctivitis.

SUMMARY:
The purpose of this study is to evaluate the comfort of BEPREVE compared to LASTACAFT after instillation.

DETAILED DESCRIPTION:
After one drop is instilled subjects will complete a comfort assessment at 1, 3, 5, and 10 minutes after drop instillation.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet the following criteria to be enrolled in this study:

1. Are male or female at least 18 years of age who are diagnosed with allergic conjunctivitis.
2. Have allergic ocular symptoms within the last three days.
3. Are willing/able to follow instructions from the study investigator and his/her staff.
4. Have signed informed consent approved by Institutional Review Board or Independent Ethics Committee.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study:

1. Have known hypersensitivity to either BEPREVE™ or LASTACAFT® or to any component of the test article (including "procedural" medications such as anesthetic and/or fluorescein drops, dilating drops, etc.).
2. Have active corneal pathology noted in the study eye at the screening visit. Active corneal pathology is defined as corneal pathology that is non stable, or greater than mild, or will compromise assessment of the safety or efficacy of treatment.
3. Are pregnant or nursing/lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are diagnosed with allergic conjunctivitis and who meet all other inclusion/exclusion criteria will be eligible to enter the study.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2011-04; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek Cunningham, OD, Principal Investigator — Dell Laser Consultants
Locations (1):
- Derek Cunningham, Austin, Texas, United States